CLINICAL TRIAL: NCT03730350
Title: A Randomized-Controlled Trial of a Novel Perioperative Acceptance and Commitment Therapy and Clinical Hypnosis Program for Postsurgical Pain and Opioid Weaning
Brief Title: Perioperative ACT-Based Clinical Hypnosis for Opioid Weaning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jo Carroll, Research Manager, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-5441
Record Dates: First submitted 2018-10-30; First posted 2018-11-05 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Post-Surgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: This study will conduct a 2-arm (intervention vs. treatment-as-usual) pilot RCT with patients currently undergoing oncology surgery at Toronto General Hospital. This study will recruit N = 92 patients (n = 46 psychology intervention, n = 46 control). The psychology intervention will be delivered by the TPS pain psychology team, under the supervision of Transitional Pain Service lead pain psychologist Dr. Aliza Weinrib. In addition, audio recordings developed by Dr. Weinrib will be provided to patients
Masking Description: Random assignment to group will take place after baseline assessment. Patients who are randomly assigned to the clinical hypnosis group will immediately undergo their first in-person hypnosis session focused on preparing for surgery. Masking is not employed as patients will know if they are randomized to the intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental): Prior to surgery, a member of the pain psychology team will guide patients through a clinical hypnosis session aimed at preparing for surgery by reducing anxiety and introducing relaxation and self-soothing strategies that can be used after surgery for adaptive coping. They will also be provided with a recording of this hypnosis script to use at home, and it will be recommended that they listen to the recording on the two days prior to surgery. Following surgery, a clinician from the pain psychology team will visit the patient in hospital on post-operative day one or whenever they are able to be seen prior to hospital discharge, in order to guide them through a clinical hypnosis session targeted at increasing comfort and pain relief.
  Interventions: Behavioral: Clinical Hypnosis
- Standard Care (No Intervention): This control group will receive standard care pre- and post-surgery. After the completion of their one-month trial, control participants will be offered access to the hypnosis recordings, as well as an in-person hypnosis session.

INTERVENTIONS:
Behavioral: Clinical Hypnosis — Hypnosis guidance and audio tracks aimed at promoting pain relief, reducing distress and anxiety, and facilitating sleep will be provided for independent use, with daily practice recommended. Each hypnosis session will be 20-25 minutes long. The scripts for these sessions have been developed based on the clinical literature (e.g., Elkins, 2014) and are already in use with patients of the pain service.
  Arms: Hypnosis

SUMMARY:
This randomized-controlled trial (RCT) will evaluate the effectiveness of a pain psychology intervention -- consisting of a hybrid of acceptance and commitment therapy (ACT) and clinical hypnosis intervention -- in reducing opioid consumption after major surgery. Consenting patients undergoing oncology surgeries at Toronto General Hospital (TGH) will be randomly assigned to one of two groups: (1) standard care or (2) standard care plus an ACT/clinical hypnosis intervention for pain management. The hypnosis intervention will be delivered via one session with a psychotherapist prior to surgery, one session with a psychotherapist after surgery, and the provision of audio recordings to guide patients in practicing self-hypnosis. The pain psychology intervention is targeted at reducing pain, as well as pain-related anxiety, distress, sleep disturbance, and functional impairment. The primary goal of the pain psychology intervention is to help patients to feel more comfortable while using less opioid medication in the week after surgery.

DETAILED DESCRIPTION:
Hypnosis is one of the oldest strategies for the management of pain; however, interest in hypnosis as a pain management strategy has ebbed and flowed over time. Given the current concern over opioid use for pain management, non-pharmacological pain management options, such as clinical hypnosis, are being revisited. In addition, over the past twenty years, there has been a new wave of scientific investigation into the efficacy of hypnosis for acute and chronic pain. As a result of this body of evidence for the efficacy of clinical hypnosis for pain management, the American Psychological Association has recommended that clinical hypnosis be included as part of standard care for pain relief, unless an individual indicates a strong aversion to it.

Previous research has investigated the utility of clinical hypnosis for pain management in the perioperative context. Surgical patients who received adjunct hypnosis treatment had better outcomes (e.g., less pain, better mood, and less medication use) than 89% of patients who received treatment as usual, as evidenced by large effect sizes across 1624 patients from randomized and non-randomized controlled trials. A more recent meta-analysis demonstrated small to medium effects in favor of hypnosis on various post-surgical outcomes (e.g., pain, emotional distress, medication consumption, and post-surgical recovery), across 2597 patients in randomized controlled trials. Although these meta-analyses have demonstrated an association between the implementation of hypnosis interventions and an overall reduction in medication consumption, previous investigations have rarely focused specifically on reduced use of opioid medication, which is important in the context of current concerns about opioid overuse.

Furthermore, meta-analyses have indicated that dysregulation of the parasympathetic nervous system is associated with the development of chronic pain, leaving sufferers unable to regulate stress, recovery, and relaxation processes. The investigators hypothesize that the relaxation associated with the clinical hypnosis intervention will lead to activation of the parasympathetic nervous system and, accordingly, greater heart rate variability. Therefore, the investigators hypothesize that patients who are randomized to the clinical hypnosis treatment will not only use less opioid medication in the week after surgery, but will also demonstrate greater heart rate variability at one month post-surgery, which is thought to protect against the development of long-term pain.

The study's goal is to provide patients with a range of strategies that will be most helpful and efficacious in reducing suffering during the pre- and post-operative periods. A secondary goal is to deliver as much therapeutic content as possible through audio recordings in order to create a psychological intervention that requires less face-to-face contact between clinician and patient, but provides more support (e.g., patients can listen to the recordings at bedtime when the clinician would not be available on a daily basis). The use of audio recordings will conserve staffing resources, while at the same time allowing for the dissemination of pain psychology tools to more patients. Therefore, in the current study, the study aims to test the feasibility and efficacy of this approach, termed ACT-Informed Clinical Hypnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80
* Scheduled for surgical oncology procedure (i.e., thoracic, gastrointestinal, gynecologic oncology, urologic, head and neck or breast cancer surgery)

Exclusion Criteria:

* Patients with limited comprehension of English who would not be able to understand the verbal instructions for clinical hypnosis
* Patients with a known history of serious mental illness (e.g., schizophrenia and/or current PTSD)
* Patients with cognitive deficits due to dementia whose comprehension may limit benefit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Opioid Use: Measured as the morphine equivalent dosage (MED) and based on conversion methods used by doctors and nurses at the University Health Network | One Week
  The effectiveness of the intervention on opioid use will be tested using a 2 factor mixed effects linear model with group (hypnosis vs. standard care) and time (pre-surgery, one week post-surgery) as factors. The investigators predict significantly lower mean daily morphine-equivalent opioid use in the hypnosis group compared to standard care at one week post surgery.
  MED values typically range between 0-200 milligrams/day and higher values mean greater opioid use.

SECONDARY OUTCOMES:
Post-Surgical Pain Intensity: Measured using the numeric rating scale (0 = no pain; 10 = most pain imaginable) | One Week
  Post-surgical pain intensity will be tested with a linear mixed effects model (group x time).
Post-Surgical Pain Interference: Measured using the Brief Pain Inventory | One Week
  Pain interference will be tested with a linear mixed effects model (group x time).
  Pain interference has seven subscales of general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. Each subscale has five likert-type response options (not at all; extremely). Pain interference will be measured as the mean ratings of the seven subscales.
Sleep Impairment; Measured using the Patient Report Outcomes Measurement Information System (PROMIS) - Sleep Disturbance and Sleep-Related Impairment | One Week
  Sleep impairment will be tested with a linear mixed effects model (group x time).
  The majority of the PROMIS items employ response scales with five options: 1 = Not at all, 2 = A little bit, 3 = Somewhat, 4 = Quite a bit, 5 = Very much.Scores are calculated from the total of item responses, with higher scores reflecting greater sleep disturbance/impairment
Mood: Measured using the Center for Epidemiological Studies Depression Scale Short-Form | One Week
  Mood symptoms will be tested with a linear mixed effect models (group x time).
  The total score is calculated by the sum of the items with higher scores reflecting greater depressive symptomatology.
Anxiety: Measured using the Generalized Anxiety Disorder Assessment | One Week
  Anxiety symptoms will be tested with a linear mixed effect models (group x time).
  This 7-item scale assesses signs of GAD (e.g. "Feeling afraid as if something awful might happen") with response options of: (1) Not at all, (2) Several days, (3) More than half the days, (4) Nearly every day. Scores are calculated from the total of item responses, with higher scores reflecting greater anxiety.
Parasympathetic Tone and Activation: Assessed by metrics of heart-rate variability (HRV) | One Month
  Parasympathetic tone and activation will be measured during conditions of resting (5 minutes) and audio-guided relaxation (10 minutes). Higher HRV values reflect greater parasympathetic tone and activation. The effects of the intervention on parasympathetic tone and activation will be tested with a linear mixed effects model with group (hypnosis, standard care) and time (pre-surgery, one month post-surgery) as between-group factors, condition (rest, relaxation) as the within-subject factor, and heart-rate variability as the dependent variable.

CONTACTS AND LOCATIONS:
Overall Officials: Hance Clarke, MD, PhD, Principal Investigator — Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jensen MP. Hypnosis for chronic pain management: a new hope. Pain. 2009 Dec;146(3):235-237. doi: 10.1016/j.pain.2009.06.027. Epub 2009 Jul 10. No abstract available. PMID 19596518
- [Background] American Psychological Association, D., Society of Psychological Hypnosis. (2004). Hypnosis for the Relief and Control of Pain. Retrieved from http://www.apa.org/research/action/hypnosis.aspx
- [Background] Koenig J, Falvay D, Clamor A, Wagner J, Jarczok MN, Ellis RJ, Weber C, Thayer JF. Pneumogastric (Vagus) Nerve Activity Indexed by Heart Rate Variability in Chronic Pain Patients Compared to Healthy Controls: A Systematic Review and Meta-Analysis. Pain Physician. 2016 Jan;19(1):E55-78. PMID 26752494
- [Derived] Azam MA, Weinrib AZ, Slepian PM, Rosenbloom BN, Waisman A, Clarke H, Katz J. Effects of perioperative clinical hypnosis on heart rate variability in patients undergoing oncologic surgery: secondary outcomes of a randomized controlled trial. Front Pain Res (Lausanne). 2024 Mar 8;5:1354015. doi: 10.3389/fpain.2024.1354015. eCollection 2024. PMID 38524266